CLINICAL TRIAL: NCT07021378
Title: Tolerance to Immunomodulatory Nutritional Therapy in Oncology Patients Undergoing Chemotherapy and Radiotherapy
Acronym: NESTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Principal Investigator, Camila Motta Venchiarutti Moniz, Doctor, Principal Investigator, D'Or Institute for Research and Education
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 55651522.2.1001.0087
Record Dates: First submitted 2025-03-31; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-10

CONDITIONS: Nutritional Deficiency; Breast Cancer; Anal Cancer
MeSH Terms: conditions — Malnutrition; Breast Neoplasms; Anus Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Pilot study to evaluate the tolerance of imune nutritional supplement during cancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: patients with HER2-positive breast cancer with dietary supplementary (Experimental): Supplementation with impact (Nestlé) and sachets to ingest during the neoadjuvant period, weeks after surgery, and adjuvant treatment.
  Interventions: Dietary Supplement: Dietary Supplement
- Control cohort A: Routine nutrition orientation (Other): Control Cohort A: According to the institutional routine nutritional orientation
  Interventions: Other: Control Cohort A
- Cohort B: Patients with anal canal cancer with dietary supplementary (Experimental): Impact supplement (Nestlé) and sachets of the supplement to ingest during chemotherapy and radiotherapy
  Interventions: Dietary Supplement: Dietary Supplement
- Control cohort B: Routine nutrition orientation (Other): Control cohort B: According to the institutional routine nutritional orientation
  Interventions: Other: Control cohort B

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Phase 1 (Neoadjuvant Chemotherapy):
  Patients will receive 2 units of Impact oral supplement and 1 sachet of protein module daily, for 7 days prior to each chemotherapy cycle.
  During the interval between the end of one cycle and 7 days before the next, 2 sachets of protein module per day will be maintained.
  Phase 2 (Surgery):
  2 units of Impact once daily, for 7 days prior to surgery.
  Phase 3 (Radiotherapy):
  2 units of Impact and 1 sachet of protein module daily, for 7 days prior to starting radiotherapy (RT), followed by 1 unit of Impact once daily throughout the course of RT.
  Protein module: 13 g/day until the end of treatment.
  Arms: Cohort A: patients with HER2-positive breast cancer with dietary supplementary
Dietary Supplement: Dietary Supplement — 2 units of Impact oral supplement and 1 sachet of protein module once daily, starting 1 week before the initiation of radiotherapy (RT).
  During RT: 1 unit of Impact and 1 sachet of protein module daily, until 1 week before the end of RT.
  2 units of Impact and 1 sachet of protein module daily until the end of treatment, starting from 1 week before the end of RT.
  Protein module: 13 g/day throughout the entire treatment period.
  Arms: Cohort B: Patients with anal canal cancer with dietary supplementary
Other: Control Cohort A — Control cohort A: According to the institutional routine nutritional orientation
  Arms: Control cohort A: Routine nutrition orientation
Other: Control cohort B — Control cohort B: According to the institutional routine nutritional orientation
  Arms: Control cohort B: Routine nutrition orientation

SUMMARY:
The importance of nutritional support is established in some types of neoplasms, especially those involving the digestive tract. Recently, nutritional supplements containing substances with proposed immunomodulatory action have been developed. It is still unclear whether the use of immunomodulatory supplements can reduce the occurrence of treatment-related toxicities in oncology, such as radiodermatitis and mucositis. The aim of this study is to investigate whether the use of supplements with immunomodulatory action could reduce the occurrence of cutaneous and mucosal toxicities in oncology treatment, such as radiodermatitis and diarrhea.

DETAILED DESCRIPTION:
A prospective pilot study will be conducted to assess the use of immunomodulatory nutritional therapy in patients undergoing chemotherapy and radiotherapy for adjuvant or definitive cancer treatment at a service affiliated with Oncologia D'Or or at the Instituto do Câncer do Estado de São Paulo.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of carcinoma from one of the following two primary sites: breast (Cohort A); anal canal (Cohort B);
2. Localized disease, stages I-III, according to the 8th edition of TNM classification;
3. Indication for neoadjuvant TC-HP treatment, surgery, and adjuvant radiotherapy for breast cancer (Cohort A) or definitive chemoradiotherapy for anal canal cancer (Cohort B).

Exclusion Criteria:

1. Metastatic disease;
2. Inability to intake food orally;
3. Conditions that compromise the ability to ingest or absorb nutritional therapy, such as inflammatory bowel disease, intestinal perforation, intestinal obstruction, or uncontrolled lower gastrointestinal bleeding;
4. Previous radiotherapy in the same field where the current treatment will be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the immunomodulatory nutritional supplementation regimen | Up to 36 weeks
  Percentage of adherence to the immunomodulatory nutritional supplementation regimen

CONTACTS AND LOCATIONS:
Overall Officials: Camila M. V. Moniz, MD-PhD, Principal Investigator — PI
Locations (2):
- Brazil (2):
  - Instituto D'or de Pesquisa e Ensino, São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Scientific dissemination - articles and conferences.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 4 years

REFERENCES:
- [Background] Colasanto JM, Prasad P, Nash MA, Decker RH, Wilson LD. Nutritional support of patients undergoing radiation therapy for head and neck cancer. Oncology (Williston Park). 2005 Mar;19(3):371-9; discussion 380-2, 387. PMID 15828552
- [Background] Jordan T, Mastnak DM, Palamar N, Kozjek NR. Nutritional Therapy for Patients with Esophageal Cancer. Nutr Cancer. 2018 Jan;70(1):23-29. doi: 10.1080/01635581.2017.1374417. Epub 2017 Oct 10. PMID 29016197
- [Background] Mileo AM, Nistico P, Miccadei S. Polyphenols: Immunomodulatory and Therapeutic Implication in Colorectal Cancer. Front Immunol. 2019 Apr 11;10:729. doi: 10.3389/fimmu.2019.00729. eCollection 2019. PMID 31031748
- [Background] van Ramshorst MS, van der Voort A, van Werkhoven ED, Mandjes IA, Kemper I, Dezentje VO, Oving IM, Honkoop AH, Tick LW, van de Wouw AJ, Mandigers CM, van Warmerdam LJ, Wesseling J, Vrancken Peeters MT, Linn SC, Sonke GS; Dutch Breast Cancer Research Group (BOOG). Neoadjuvant chemotherapy with or without anthracyclines in the presence of dual HER2 blockade for HER2-positive breast cancer (TRAIN-2): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2018 Dec;19(12):1630-1640. doi: 10.1016/S1470-2045(18)30570-9. Epub 2018 Nov 6. PMID 30413379
- [Background] Boisselier P, Kaminsky MC, Thezenas S, Gallocher O, Lavau-Denes S, Garcia-Ramirez M, Alfonsi M, Cupissol D, de Forges H, Janiszewski C, Geoffrois L, Sire C, Senesse P; Head and Neck Oncology and Radiotherapy Group (GORTEC). A double-blind phase III trial of immunomodulating nutritional formula during adjuvant chemoradiotherapy in head and neck cancer patients: IMPATOX. Am J Clin Nutr. 2020 Dec 10;112(6):1523-1531. doi: 10.1093/ajcn/nqaa227. PMID 32936874
- [Background] Talvas J, Garrait G, Goncalves-Mendes N, Rouanet J, Vergnaud-Gauduchon J, Kwiatkowski F, Bachmann P, Bouteloup C, Bienvenu J, Vasson MP. Immunonutrition stimulates immune functions and antioxidant defense capacities of leukocytes in radiochemotherapy-treated head & neck and esophageal cancer patients: A double-blind randomized clinical trial. Clin Nutr. 2015 Oct;34(5):810-7. doi: 10.1016/j.clnu.2014.12.002. Epub 2014 Dec 9. PMID 25575640